CLINICAL TRIAL: NCT04930471
Title: A Multi-center, Prospective, Cohort Study to Elucidate the Effects of Metformin Treatment on Steroid Hormones and Social Behavior. Linking Autistic Behaviorial Symptoms to Changes in Steroid Hormone Availability
Brief Title: Steroid and Behaviour Changes Under Metformin
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Lindenhofstiftung (Unknown)
Responsible Party: Sponsor
Other Study IDs: Steroid Changes Metformin
Record Dates: First submitted 2021-06-01; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Autistic Disorder
Keywords: Steroid hormones; GC-MS; urine analysis; androgens; autism spectrum disorders
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Metformin (all participants): Patients with a new indication for Metformin (standard dosage as assigned by the treating physician) therapy. Samples will be collected before and after 12 weeks of Metformin treatment.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Treatment with Metformin as prescribed by the treating physician.

SUMMARY:
Background

Based on various suggestions, social behavior is mediated by a change in steroid hormones. These have diverse effects on the (neuro-)development during critical stages, whereby especially androgen and insulin metabolism seem to play a key role. Various lines of evidence indicate that metformin could influence and improve the symptoms of social withdrawal. Therefore, the investigators will analyze urinary samples of patients before and after treatment with metformin to elucidate the changes in steroid hormone profiles and measure changes in social behavior to examine a potential correlation.

Material & Methods

Steroid hormone analysis including the most prominent androgen, estrogen, progesterone, aldosterone, corticosterone, cortisone and cortisol metabolites analyzed with gas chromatography mass spectrometry and a questionnaire (Autism-Spectrum Quotient) will be performed prior to and after 12-weeks metformin treatment.

Discussion

It is likely, that due to different pathophysiological mechanisms such as an effect on respiratory chain in mitochondria or via AMP activated protein kinase a general reduction of total androgens will be detected prior versus post metformin treatment. The encompassing measurement of steroid hormones will allow to detect influences on different metabolites and in consequence enzyme activities. The potential changes prior versus post shall give hints concerning the involvement of specific cascades involved, with potential pharmacological targets for future research.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus and an indication for metformin according to the American Diabetes Association (American Diabetes Association, 2021a) starting a new metformin treatment. The main marker will be fasting plasma glucose levels of 7.0mmol/L and/or HbA1c 6.5% (American Diabetes Association, 2021a).
* Written informed consent.

Exclusion Criteria:

* Patients under 18 years of age.
* Clinically significant concomitant disease (e.g. advanced renal failure, hepatic dysfunction, neoplasia).
* Significant musculoskeletal disease.
* Active infection during sample collection.
* Immunosuppressive medical therapy.
* Hormonal/steroid treatment.
* Pregnancy.
* Psychiatric disease and known social behavior altering medication (e.g. antipsychotic medication).
* Known or suspected malcompliance, drug or alcohol abuse.
* Inability to follow the procedures of the study, e.g. due to insufficient language skills, severe dementia.
* Life-expectancy < 6 months.
* Poor tolerability to metformin treatment with following treatment discontinuation within duration of follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the the Lindenhofgruppe and its associated practices with a new indication for Metformin treatment.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Changes in GC-MS measured urinary androgen metabolite levels. | After 12 weeks follow-up
  Changes in urinary androgen metabolite levels of interest (see below) prior to metformin treatment start and after 12-weeks of treatment.
  Hormones of interest include Androgen-Metabolites (Androsterone, Androstenediol, 11-Oxoetiocholanolone, 11β-Hydroxyandrosterone, 11β-Hydroxyetiocholanolone, Dehydroepiandrosterone, 5-Androstene-3β,17β-diol, 16α-Hydroxydehydroepiandrosterone, 5-Androstene-3β,16α,17β-triol, 5-Pregnene-3β, 16α,17β-triol, Testosterone, 5α-Dihydrotestosterone). All will be measured in urinary samples using GC-MS (gas-chromatography mass-spectrometry).
Changes in GC-MS measured urinary oestrogen metabolite levels. | After 12 weeks follow-up
  Changes in urinary oestrogen metabolite levels of interest (see below) prior to metformin treatment start and after 12-weeks of treatment.
  Hormones of interest include Oestrogen-Metabolites (Estriol, 17b-Estradiol), Progesterone-Metabolites (17-Hydroxypregnanolone, Pregnanediol, Pregnanetriol, 11-Oxo-Pregnanetriol). All wil be measured in urinary samples using GC-MS (gas-chromatography mass-spectrometry).
Changes in GC-MS measured urinary progesterone metabolite levels. | After 12 weeks follow-up
  Changes in urinary progesterone metabolite levels of interest (see below) prior to metformin treatment start and after 12-weeks of treatment.
  Hormones of interest include Progesterone-Metabolites (17-Hydroxypregnanolone, Pregnanediol, Pregnanetriol, 11-Oxo-Pregnanetriol).
  All wil be measured in urinary samples using GC-MS (gas-chromatography mass-spectrometry).
Changes in GC-MS measured urinary aldosterone metabolite levels. | After 12 weeks follow-up
  Changes in urinary aldosterone metabolite levels of interest (see below) prior to metformin treatment start and after 12-weeks of treatment.
  Hormones of interest include Aldosterone-Metabolites (Tetrahydroaldosterone). All wil be measured in urinary samples using GC-MS (gas-chromatography mass-spectrometry).
Changes in GC-MS measured urinary corticosterone metabolite levels. | After 12 weeks follow-up
  Changes in urinary corticosterone metabolite levels of interest (see below) prior to metformin treatment start and after 12-weeks of treatment.
  Hormones of interest include Corticosterone-Metabolites (TetrahydroDOC, Tetrahydrodehydrocorticosterone, Tetrahydrocorticosterone, 5a-Tetrahydrocorticosterone, 18-Hydroxy-tetrahydrocompound A, Cortisone).
  All wil be measured in urinary samples using GC-MS (gas-chromatography mass-spectrometry).
Changes in GC-MS measured urinary cortisone metabolite levels. | After 12 weeks follow-up
  Changes in urinary cortisone metabolite levels of interest (see below) prior to metformin treatment start and after 12-weeks of treatment.
  Hormones of interest include Cortisone-Metabolites (Tetrahydrocortisone, a-Cortolone, b-Cortolone, 20a-Dihydrocortisone, 20b-Dihydrocortisone).
  All wil be measured in urinary samples using GC-MS (gas-chromatography mass-spectrometry).
Changes in GC-MS measured urinary cortisol metabolite levels. | After 12 weeks follow-up
  Changes in urinary cortisol metabolite levels of interest (see below) prior to metformin treatment start and after 12-weeks of treatment.
  Hormones of interest include Cortisol-Metabolites (Cortisol, Tetrahydrocortisol, 5a-Tetrahydrocortisol, a-Cortol, b-Cortol, 20a-Dihydrocortisol, 6b-Hydroxycortisol, 18-Hydroxycortisol).
  All wil be measured in urinary samples using GC-MS (gas-chromatography mass-spectrometry).
Behavioral Changes | After 12 weeks follow-up
  Changes in social behavior measured by the Autism-Spectrum Quotient AQ prior to metformin treatment start and after 12-weeks of treatment.

SECONDARY OUTCOMES:
Correlation between urinary steroid hormone level changes (metabolites of androgen, oestrogen, progesterone, aldosterone, corticosterone, cortisone and cortisol) and behavioral changes measured with pearson correlation coefficient. | After 12 weeks follow-up
  A potential correlation and/or dosage effect between the primary outcomes will be evaluated using the pearson correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Markus G Mohaupt, Professor, Study Director — Lindenhofgruppe Berne and Inselspital Berne, Department of Nephrology
Locations (1):
- Lindenhofgruppe, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andonian MR, Barrett AS, Vinogradov SN. Physical properties and subunits of Haemopis grandis erythrocruorin. Biochim Biophys Acta. 1975 Dec 15;412(2):202-13. doi: 10.1016/0005-2795(75)90035-5. PMID 84
- [Background] Aufdenblatten M, Baumann M, Raio L, Dick B, Frey BM, Schneider H, Surbek D, Hocher B, Mohaupt MG. Prematurity is related to high placental cortisol in preeclampsia. Pediatr Res. 2009 Feb;65(2):198-202. doi: 10.1203/PDR.0b013e31818d6c24. PMID 19047954
- [Background] Azziz R. Androgen excess is the key element in polycystic ovary syndrome. Fertil Steril. 2003 Aug;80(2):252-4. doi: 10.1016/s0015-0282(03)00735-0. No abstract available. PMID 12909479
- [Background] Baillargeon JP, Jakubowicz DJ, Iuorno MJ, Jakubowicz S, Nestler JE. Effects of metformin and rosiglitazone, alone and in combination, in nonobese women with polycystic ovary syndrome and normal indices of insulin sensitivity. Fertil Steril. 2004 Oct;82(4):893-902. doi: 10.1016/j.fertnstert.2004.02.127. PMID 15482765
- [Background] Baron-Cohen S, Wheelwright S, Skinner R, Martin J, Clubley E. The autism-spectrum quotient (AQ): evidence from Asperger syndrome/high-functioning autism, males and females, scientists and mathematicians. J Autism Dev Disord. 2001 Feb;31(1):5-17. doi: 10.1023/a:1005653411471. PMID 11439754
- [Background] Biag HMB, Potter LA, Wilkins V, Afzal S, Rosvall A, Salcedo-Arellano MJ, Rajaratnam A, Manzano-Nunez R, Schneider A, Tassone F, Rivera SM, Hagerman RJ. Metformin treatment in young children with fragile X syndrome. Mol Genet Genomic Med. 2019 Nov;7(11):e956. doi: 10.1002/mgg3.956. Epub 2019 Sep 14. PMID 31520524
- [Background] Bishop DV, Maybery M, Maley A, Wong D, Hill W, Hallmayer J. Using self-report to identify the broad phenotype in parents of children with autistic spectrum disorders: a study using the Autism-Spectrum Quotient. J Child Psychol Psychiatry. 2004 Nov;45(8):1431-6. doi: 10.1111/j.1469-7610.2004.00849.x. PMID 15482503
- [Background] Brandt EJ, Elliott RW, Swank RT. Defective lysosomal enzyme secretion in kidneys of Chediak-Higashi (beige) mice. J Cell Biol. 1975 Dec;67(3):774-88. doi: 10.1083/jcb.67.3.774. PMID 408
- [Background] Burghen GA, Givens JR, Kitabchi AE. Correlation of hyperandrogenism with hyperinsulinism in polycystic ovarian disease. J Clin Endocrinol Metab. 1980 Jan;50(1):113-6. doi: 10.1210/jcem-50-1-113. PMID 7350174
- [Background] Campagnoli C, Abba C, Ambroggio S, Brucato T, Pasanisi P. Life-style and metformin for the prevention of endometrial pathology in postmenopausal women. Gynecol Endocrinol. 2013 Feb;29(2):119-24. doi: 10.3109/09513590.2012.706671. Epub 2012 Sep 5. PMID 22946682
- [Background] Chakrabarti B, Dudbridge F, Kent L, Wheelwright S, Hill-Cawthorne G, Allison C, Banerjee-Basu S, Baron-Cohen S. Genes related to sex steroids, neural growth, and social-emotional behavior are associated with autistic traits, empathy, and Asperger syndrome. Autism Res. 2009 Jun;2(3):157-77. doi: 10.1002/aur.80. PMID 19598235
- [Background] Chang RJ, Nakamura RM, Judd HL, Kaplan SA. Insulin resistance in nonobese patients with polycystic ovarian disease. J Clin Endocrinol Metab. 1983 Aug;57(2):356-9. doi: 10.1210/jcem-57-2-356. PMID 6223044
- [Background] Chaoui R, Bollmann R, Zienert A, Weichold K, Goldner B, Semmler K. [Prenatal diagnosis of truncus arteriosus communis (type I) in diabetic pregnancy]. Zentralbl Gynakol. 1992;114(4):198-200. German. PMID 1621459
- [Background] Chou KH, von Eye Corleta H, Capp E, Spritzer PM. Clinical, metabolic and endocrine parameters in response to metformin in obese women with polycystic ovary syndrome: a randomized, double-blind and placebo-controlled trial. Horm Metab Res. 2003 Feb;35(2):86-91. doi: 10.1055/s-2003-39056. PMID 12734787
- [Background] Cibula D, Fanta M, Vrbikova J, Stanicka S, Dvorakova K, Hill M, Skrha J, Zivny J, Skrenkova J. The effect of combination therapy with metformin and combined oral contraceptives (COC) versus COC alone on insulin sensitivity, hyperandrogenaemia, SHBG and lipids in PCOS patients. Hum Reprod. 2005 Jan;20(1):180-4. doi: 10.1093/humrep/deh588. Epub 2004 Dec 2. PMID 15576394
- [Background] El-Baz F, Hamza RT, Ayad MS, Mahmoud NH. Hyperandrogenemia in male autistic children and adolescents: relation to disease severity. Int J Adolesc Med Health. 2014;26(1):79-84. doi: 10.1515/ijamh-2012-0116. PMID 23612632
- [Background] Gambineri A, Pelusi C, Genghini S, Morselli-Labate AM, Cacciari M, Pagotto U, Pasquali R. Effect of flutamide and metformin administered alone or in combination in dieting obese women with polycystic ovary syndrome. Clin Endocrinol (Oxf). 2004 Feb;60(2):241-9. doi: 10.1111/j.1365-2265.2004.01973.x. PMID 14725687
- [Background] Gantois I, Popic J, Khoutorsky A, Sonenberg N. Metformin for Treatment of Fragile X Syndrome and Other Neurological Disorders. Annu Rev Med. 2019 Jan 27;70:167-181. doi: 10.1146/annurev-med-081117-041238. Epub 2018 Oct 26. PMID 30365357
- [Background] Garfunkel D, Anagnostou EA, Aman MG, Handen BL, Sanders KB, Macklin EA, Chan J, Veenstra-VanderWeele J. Pharmacogenetics of Metformin for Medication-Induced Weight Gain in Autism Spectrum Disorder. J Child Adolesc Psychopharmacol. 2019 Aug;29(6):448-455. doi: 10.1089/cap.2018.0171. Epub 2019 Jun 12. PMID 31188026
- [Background] Gasser BA, Kurz J, Dick B, Mohaupt MG. A reply to 'Alteration of steroidogenesis in boys with autism spectrum disorders'. Transl Psychiatry. 2021 May 10;11(1):278. doi: 10.1038/s41398-021-01393-9. No abstract available. PMID 33972510
- [Background] Gasser BA, Kurz J, Dick B, Mohaupt MG. Steroid Metabolites Support Evidence of Autism as a Spectrum. Behav Sci (Basel). 2019 May 9;9(5):52. doi: 10.3390/bs9050052. PMID 31075898
- [Background] Gasser BA, Kurz J, Dick B, Mohaupt MG. Are Steroid Hormones Dysregulated in Autistic Girls? Diseases. 2020 Mar 14;8(1):6. doi: 10.3390/diseases8010006. PMID 32183287
- [Background] Gasser BA, Kurz J, Senn W, Escher G, Mohaupt MG. Stress-induced alterations of social behavior are reversible by antagonism of steroid hormones in C57/BL6 mice. Naunyn Schmiedebergs Arch Pharmacol. 2021 Jan;394(1):127-135. doi: 10.1007/s00210-020-01970-7. Epub 2020 Sep 7. PMID 32894324
- [Background] Hirsch A, Hahn D, Kempna P, Hofer G, Nuoffer JM, Mullis PE, Fluck CE. Metformin inhibits human androgen production by regulating steroidogenic enzymes HSD3B2 and CYP17A1 and complex I activity of the respiratory chain. Endocrinology. 2012 Sep;153(9):4354-66. doi: 10.1210/en.2012-1145. Epub 2012 Jul 9. PMID 22778212
- [Background] Ibanez L, Valls C, Marcos MV, Ong K, Dunger DB, De Zegher F. Insulin sensitization for girls with precocious pubarche and with risk for polycystic ovary syndrome: effects of prepubertal initiation and postpubertal discontinuation of metformin treatment. J Clin Endocrinol Metab. 2004 Sep;89(9):4331-7. doi: 10.1210/jc.2004-0463. PMID 15356029
- [Background] Ingudomnukul E, Baron-Cohen S, Wheelwright S, Knickmeyer R. Elevated rates of testosterone-related disorders in women with autism spectrum conditions. Horm Behav. 2007 May;51(5):597-604. doi: 10.1016/j.yhbeh.2007.02.001. Epub 2007 Feb 8. PMID 17462645
- [Background] Ito-Yamaguchi A, Suganuma R, Kumagami A, Hashimoto S, Yoshida-Komiya H, Fujimori K. Effects of metformin on endocrine, metabolic milieus and endometrial expression of androgen receptor in patients with polycystic ovary syndrome. Gynecol Endocrinol. 2015 Jan;31(1):44-7. doi: 10.3109/09513590.2014.951321. Epub 2014 Sep 19. PMID 25237893
- [Background] Jansakova K, Hill M, Celarova D, Celusakova H, Repiska G, Bicikova M, Macova L, Ostatnikova D. Alteration of the steroidogenesis in boys with autism spectrum disorders. Transl Psychiatry. 2020 Oct 6;10(1):340. doi: 10.1038/s41398-020-01017-8. PMID 33024080
- [Background] Kaji A, Saheki T. Endo-arabinanase from Bacillus subtilis F-11. Biochim Biophys Acta. 1975 Dec 18;410(2):354-60. doi: 10.1016/0005-2744(75)90237-5. PMID 1096
- [Background] Kempna P, Marti N, Udhane S, Fluck CE. Regulation of androgen biosynthesis - A short review and preliminary results from the hyperandrogenic starvation NCI-H295R cell model. Mol Cell Endocrinol. 2015 Jun 15;408:124-32. doi: 10.1016/j.mce.2014.12.015. Epub 2014 Dec 24. PMID 25543021
- [Background] King P, Peacock I, Donnelly R. The UK prospective diabetes study (UKPDS): clinical and therapeutic implications for type 2 diabetes. Br J Clin Pharmacol. 1999 Nov;48(5):643-8. doi: 10.1046/j.1365-2125.1999.00092.x. No abstract available. PMID 10594464
- [Background] Knickmeyer R, Baron-Cohen S, Fane BA, Wheelwright S, Mathews GA, Conway GS, Brook CG, Hines M. Androgens and autistic traits: A study of individuals with congenital adrenal hyperplasia. Horm Behav. 2006 Jun;50(1):148-53. doi: 10.1016/j.yhbeh.2006.02.006. Epub 2006 Apr 19. PMID 16624315
- [Background] Kuhla A, Brichmann E, Ruhlmann C, Thiele R, Meuth L, Vollmar B. Metformin Therapy Aggravates Neurodegenerative Processes in ApoE-/- Mice. J Alzheimers Dis. 2019;68(4):1415-1427. doi: 10.3233/JAD-181017. PMID 30909226
- [Background] Lundberg IE, Nader GA. Molecular effects of exercise in patients with inflammatory rheumatic disease. Nat Clin Pract Rheumatol. 2008 Nov;4(11):597-604. doi: 10.1038/ncprheum0929. Epub 2008 Oct 7. PMID 18839010
- [Background] Luo F, Das A, Chen J, Wu P, Li X, Fang Z. Metformin in patients with and without diabetes: a paradigm shift in cardiovascular disease management. Cardiovasc Diabetol. 2019 Apr 27;18(1):54. doi: 10.1186/s12933-019-0860-y. PMID 31029144
- [Background] Majewska MD, Hill M, Urbanowicz E, Rok-Bujko P, Bienkowski P, Namyslowska I, Mierzejewski P. Marked elevation of adrenal steroids, especially androgens, in saliva of prepubertal autistic children. Eur Child Adolesc Psychiatry. 2014 Jun;23(6):485-98. doi: 10.1007/s00787-013-0472-0. Epub 2013 Sep 17. PMID 24043498
- [Background] Martin-Montalvo A, Mercken EM, Mitchell SJ, Palacios HH, Mote PL, Scheibye-Knudsen M, Gomes AP, Ward TM, Minor RK, Blouin MJ, Schwab M, Pollak M, Zhang Y, Yu Y, Becker KG, Bohr VA, Ingram DK, Sinclair DA, Wolf NS, Spindler SR, Bernier M, de Cabo R. Metformin improves healthspan and lifespan in mice. Nat Commun. 2013;4:2192. doi: 10.1038/ncomms3192. PMID 23900241
- [Background] Mathur N, Pedersen BK. Exercise as a mean to control low-grade systemic inflammation. Mediators Inflamm. 2008;2008:109502. doi: 10.1155/2008/109502. Epub 2009 Jan 11. PMID 19148295
- [Background] Misugi T, Ozaki K, El Beltagy K, Tokuyama O, Honda K, Ishiko O. Insulin-lowering agents inhibit synthesis of testosterone in ovaries of DHEA-induced PCOS rats. Gynecol Obstet Invest. 2006;61(4):208-15. doi: 10.1159/000091496. Epub 2006 Feb 13. PMID 16479139
- [Background] Morin-Papunen L, Vauhkonen I, Koivunen R, Ruokonen A, Martikainen H, Tapanainen JS. Metformin versus ethinyl estradiol-cyproterone acetate in the treatment of nonobese women with polycystic ovary syndrome: a randomized study. J Clin Endocrinol Metab. 2003 Jan;88(1):148-56. doi: 10.1210/jc.2002-020997. PMID 12519844
- [Background] Nestler JE, Jakubowicz DJ. Lean women with polycystic ovary syndrome respond to insulin reduction with decreases in ovarian P450c17 alpha activity and serum androgens. J Clin Endocrinol Metab. 1997 Dec;82(12):4075-9. doi: 10.1210/jcem.82.12.4431. PMID 9398716
- [Background] Pangrazzi L, Balasco L, Bozzi Y. Natural Antioxidants: A Novel Therapeutic Approach to Autism Spectrum Disorders? Antioxidants (Basel). 2020 Nov 26;9(12):1186. doi: 10.3390/antiox9121186. PMID 33256243
- [Background] Pedersen BK, Saltin B. Evidence for prescribing exercise as therapy in chronic disease. Scand J Med Sci Sports. 2006 Feb;16 Suppl 1:3-63. doi: 10.1111/j.1600-0838.2006.00520.x. PMID 16451303
- [Background] Protic D, Aydin EY, Tassone F, Tan MM, Hagerman RJ, Schneider A. Cognitive and behavioral improvement in adults with fragile X syndrome treated with metformin-two cases. Mol Genet Genomic Med. 2019 Jul;7(7):e00745. doi: 10.1002/mgg3.745. Epub 2019 May 18. PMID 31104364
- [Background] Rossignol DA, Frye RE. Evidence linking oxidative stress, mitochondrial dysfunction, and inflammation in the brain of individuals with autism. Front Physiol. 2014 Apr 22;5:150. doi: 10.3389/fphys.2014.00150. eCollection 2014. PMID 24795645
- [Background] Ruddy RM, Adams KV, Morshead CM. Age- and sex-dependent effects of metformin on neural precursor cells and cognitive recovery in a model of neonatal stroke. Sci Adv. 2019 Sep 11;5(9):eaax1912. doi: 10.1126/sciadv.aax1912. eCollection 2019 Sep. PMID 31535024
- [Background] Ruta L, Ingudomnukul E, Taylor K, Chakrabarti B, Baron-Cohen S. Increased serum androstenedione in adults with autism spectrum conditions. Psychoneuroendocrinology. 2011 Sep;36(8):1154-63. doi: 10.1016/j.psyneuen.2011.02.007. Epub 2011 Mar 12. PMID 21398041
- [Background] Schwarz E, Guest PC, Rahmoune H, Wang L, Levin Y, Ingudomnukul E, Ruta L, Kent L, Spain M, Baron-Cohen S, Bahn S. Sex-specific serum biomarker patterns in adults with Asperger's syndrome. Mol Psychiatry. 2011 Dec;16(12):1213-20. doi: 10.1038/mp.2010.102. Epub 2010 Sep 28. PMID 20877284
- [Background] Shackleton CH. Profiling steroid hormones and urinary steroids. J Chromatogr. 1986 Jun 20;379:91-156. doi: 10.1016/s0378-4347(00)80683-0. PMID 3525596
- [Background] Takagishi H, Takahashi T, Yamagishi T, Shinada M, Inukai K, Tanida S, Mifune N, Horita Y, Hashimoto H, Yang Y, Kameda T. Salivary testosterone levels and autism-spectrum quotient in adults. Neuro Endocrinol Lett. 2010;31(6):837-41. PMID 21196912
- [Background] Tan X, Li S, Chang Y, Fang C, Liu H, Zhang X, Wang Y. Effect of metformin treatment during pregnancy on women with PCOS: a systematic review and meta-analysis. Clin Invest Med. 2016 Sep 11;39(4):E120-31. doi: 10.25011/cim.v39i4.27091. PMID 27619399
- [Background] Tang T, Glanville J, Hayden CJ, White D, Barth JH, Balen AH. Combined lifestyle modification and metformin in obese patients with polycystic ovary syndrome. A randomized, placebo-controlled, double-blind multicentre study. Hum Reprod. 2006 Jan;21(1):80-9. doi: 10.1093/humrep/dei311. Epub 2005 Sep 30. PMID 16199429
- [Background] Tordjman S, Anderson GM, McBride PA, Hertzig ME, Snow ME, Hall LM, Ferrari P, Cohen DJ. Plasma androgens in autism. J Autism Dev Disord. 1995 Jun;25(3):295-304. doi: 10.1007/BF02179290. PMID 7559294
- [Background] Viollet B, Guigas B, Sanz Garcia N, Leclerc J, Foretz M, Andreelli F. Cellular and molecular mechanisms of metformin: an overview. Clin Sci (Lond). 2012 Mar;122(6):253-70. doi: 10.1042/CS20110386. PMID 22117616
- [Background] Wang Y, Liu B, Yang Y, Wang Y, Zhao Z, Miao Z, Zhu J. Metformin exerts antidepressant effects by regulated DNA hydroxymethylation. Epigenomics. 2019 May;11(6):655-667. doi: 10.2217/epi-2018-0187. Epub 2019 Feb 13. PMID 30760033
- [Background] Woodbury-Smith MR, Robinson J, Wheelwright S, Baron-Cohen S. Screening adults for Asperger Syndrome using the AQ: a preliminary study of its diagnostic validity in clinical practice. J Autism Dev Disord. 2005 Jun;35(3):331-5. doi: 10.1007/s10803-005-3300-7. PMID 16119474
- [Background] Xu Y, Wu Y, Huang Q. Comparison of the effect between pioglitazone and metformin in treating patients with PCOS:a meta-analysis. Arch Gynecol Obstet. 2017 Oct;296(4):661-677. doi: 10.1007/s00404-017-4480-z. Epub 2017 Aug 2. PMID 28770353
- [Background] Zemdegs J, Martin H, Pintana H, Bullich S, Manta S, Marques MA, Moro C, Laye S, Ducrocq F, Chattipakorn N, Chattipakorn SC, Rampon C, Penicaud L, Fioramonti X, Guiard BP. Metformin Promotes Anxiolytic and Antidepressant-Like Responses in Insulin-Resistant Mice by Decreasing Circulating Branched-Chain Amino Acids. J Neurosci. 2019 Jul 24;39(30):5935-5948. doi: 10.1523/JNEUROSCI.2904-18.2019. Epub 2019 Jun 3. PMID 31160539
- [Background] Zhou J, Massey S, Story D, Li L. Metformin: An Old Drug with New Applications. Int J Mol Sci. 2018 Sep 21;19(10):2863. doi: 10.3390/ijms19102863. PMID 30241400
- [Background] Zhu W, Han B, Fan M, Wang N, Wang H, Zhu H, Cheng T, Zhao S, Song H, Qiao J. Oxidative stress increases the 17,20-lyase-catalyzing activity of adrenal P450c17 through p38alpha in the development of hyperandrogenism. Mol Cell Endocrinol. 2019 Mar 15;484:25-33. doi: 10.1016/j.mce.2019.01.020. Epub 2019 Jan 23. PMID 30682387